CLINICAL TRIAL: NCT03932292
Title: Prospective Comparator Study to Evaluate the Efficacy and Tolerability of Ectoin® Mouth Wash (EML03) in the Prevention and Treatment of Radiation-induced Oral Mucositis
Brief Title: Ectoin® Mouth Wash (EML03) in the Prevention and Treatment of Radiation-induced Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: btph-002-2018-EML03
Record Dates: First submitted 2019-04-17; First posted 2019-04-30 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Oral Mucositis Due to Radiation
Keywords: Ectoin; Oral mucositis; Radiotherapy; Medical Device; Non interventional study; Mouth Wash; §23b Medical Device Act
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ectoin Mouth Wash (Active Comparator): 30 patients obtaining EML03 treatment
  Interventions: Drug: Ectoin Mouth Wash
- Supersaturated solution of calcium and phosphate ions (Active Comparator): 20 patients taking standard treatment (calcium phosphate mouth wash)
  Interventions: Drug: Supersaturated solution of calcium and phosphate ions

INTERVENTIONS:
Drug: Ectoin Mouth Wash — According to medical prescription of the instruction for use under consideration (at least 4x1 ampoule (5ml) daily, rinsed in the mouth for at least 30 seconds)
  Arms: Ectoin Mouth Wash
Drug: Supersaturated solution of calcium and phosphate ions — According to medical prescription of the instruction for use under consideration (4 times a day).
  Arms: Supersaturated solution of calcium and phosphate ions

SUMMARY:
This prospective non-interventional comparator study is to collect data on the clinical effectiveness and compliance of Ectoin® Mouth Wash solution (EML03) and to proof superiority to a well-established medical device on the market in the prevention of radiation-induced mucositis. The study doesn´t intervene with routine treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals regardless of gender older than 18 years
* Patients diagnosed with squamous cell carcinomas [SCCHN] without metastases of other nonhead and nonneck tumors
* Patients receiving radiotherapy with a Karnofsky performance index >70%
* Absence of any sign of oral mucositis at baseline (visit 1)
* A definitive or postoperative treatment
* Radiation therapy dosage: Limitation dose rate of 60-70 Gy
* Radiotherapy of 6-7 weeks duration

Exclusion Criteria:

* Subjects younger than 18 years
* Hypersensitivity to Ectoin® or any of the other ingredients of the mouth wash
* Pregnancy or breastfeeding women
* Any disease that can, in the opinion of the treating physician, affect the outcome of the observational trial
* Patients who had a history of previous radiotherapy in head-neck region or chemotherapy
* Massive alcoholic anamnesis
* Massive smoker >20 cigarettes per day at present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Change in degree of mucositis (according to WHO classification of mucositis grade) documented by the physician | Visit 1 (day 0), Visit 2 (after 14 days), Visit 3 (after 28 days), Visit 4 (after 42 days), Visit 5 (28 days after the last RT)
  The degree of oral mucositis will be assessed as follow: grade 0, no signs or symptoms; grade 1, oral soreness and erythema; grade 2, oral erythema, ulcers and solid diet tolerated; grade 3, oral ulcers and liquid diet only; grade 4, oral alimentation impossible
Change in mucositis symptoms dry mucosa, irritation of mucosa, coated tongue, unpleasant breath, decreased saliva release, pain, swelling, ulcer, difficulty to speak and difficulty to eat and dring by using a Numeric Rating Scale | day 0, day 14, day 26, day 42, Visit 5 (28 days after the last RT)
  Mucositis symptoms will be measured by using a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms).

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events will be assessed by using the Suspect Adverse Reaction Report Form (CIOMS Form I) | within 28 days after starting radiotherapy
  All occuring adverse events/serious adverse events will be documented during the entire study period.
Changes in Karnofsky status over time by using the Karnofsky Performance Scale (KPS) | Visit 1 (day 0), Visit 2 (after 14 days), Visit 3 (after 28 days), Visit 4 (after 42 days), Visit 5 (after 28 days after the last RT)
  The KPS index allows patients to be classified as to their functional impairment and describes a patient's functional status as a comprehensive 11-point scale correlating to percentage values ranging from 100% (no symptoms) to 0% (death).
Tolerability assessment by using a subsequent patient questionnaire | day 28
  The following score system will be used to quantify these evaluation: "very good" = 4; "good" =3; "neither good nor bad" = 2; "bad" = 1 and "very bad" = 0.
Satisfaction assessed by a subsequent patient questionnaire | day 28
  The following score system will be used to quantify these evaluation: "yes" 2; "maybe" = 1; and "no" = 0.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bilstein, PhD, Study Chair — Bitop AG
Locations (1):
- Department of Radiotherapy, National Institute of Oncology, Budapest, Hungary